CLINICAL TRIAL: NCT03591705
Title: Transarterial Chemoembolization Versus Transarterial Chemoembolization With Hepatic Artery Chemotherapy Infusion for Patients With Potentially Resectable HCC
Brief Title: TACE-HAIC vs. HAIC for Potentially Resectable HCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yunfei Yuan, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2018-044
Record Dates: First submitted 2018-07-09; First posted 2018-07-19 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Potentially Resection; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TACE-HAIC (Experimental): hepatic artery chemo-lipiodolization with EADM, followed by FOLFOX-based chemotherapy artery infusion
  Interventions: Drug: TACE-HAIC
- HAIC (Active Comparator): FOLFOX-based chemotherapy hepatic artery infusion
  Interventions: Drug: HAIC

INTERVENTIONS:
Drug: TACE-HAIC — transcatheter arterial chemo-lipiodolization with EADM 30mg/m2, followed by hepatic artery infusion Oxa 85 mg/m2, CF 400 mg/m2, 5-Fu 400 mg/m2, 5-Fu 1200mg/m2 infusion 23h.
  Arms: TACE-HAIC
Drug: HAIC — hepatic artery infusion Oxa 85 mg/m2, CF 400 mg/m2, 5-Fu 400 mg/m2, 5-Fu 1200mg/m2 infusion 23h.
  Arms: HAIC

SUMMARY:
Hepatocellular carcinoma (HCC) is one of the most commonly malignant tumors around the world. Hepatic resection or liver transplantation is the radical method to cure the disease. However, due to large tumors, surgical treatment is suitable for early-stage and well-reserved liver function patients. Therefore, in clinical practice, transarterial chemoembolization (TACE) is a preferential and standard treatment of potentially resectable HCC.

EACH trial opened the door to FOLFOX-based system chemotherapy for advanced HCC patients. Recently, investigators have showed that hepatic arterial infusion of FOLFOX-based chemotherapy (HAIC) was safe and efficient for HCC patients. Several clinical studies showed that HAIC bring better tumor response rate that the conditional TACE. The combination of TACE with HAIC (TACE-HAIC), theoretically can significantly increase the local doses of chemotherapeutic agents in the liver, reduce the viability of HCC cells and increase the hepatectomy rate. However, this hasn't been verified in clinical application. To identify a more effective and safety way for treating potentially resectable HCC patients, this study is designed to compare the safety and efficacy between HAIC and TACE-HAIC for those patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL)
* Diagnosed as potentially resectable with consensus by the panel of liver surgeons
* stage BCLC A/B, without extra-hepatic involvement
* No previous anti-HCC treatment
* Eastern Co-operative Group performance status 2 or less
* Liver function: Child's A or B (score < 7)

Exclusion Criteria:

* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* underlying serve cardiac or renal diseases
* Known or suspected allergy to the investigational agent or any agent given in association with this trial
* Patients ineligible for hepatic artery embolization

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2018-07-06 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 6-12 months
  Time to progression, last follow-up or death after random assignment to TACE-HAIC or HAIC

SECONDARY OUTCOMES:
overall survival | 6-12 months
  time to death or last follow-up after random assignment to TACE-HAIC or HAIC
Downstage hepatectomy rate | 6-12 months
  The hepatectomy rate after TACE-HAIC or HAIC

CONTACTS AND LOCATIONS:
Overall Officials: Yunfei Yuan, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No